CLINICAL TRIAL: NCT00180466
Title: Providing Regional Observations to Study Predictors of Events in the Coronary Tree (PROSPECT) An Imaging Study in Patients With Unstable Atherosclerotic Lesions
Brief Title: PROSPECT: An Imaging Study in Patients With Unstable Atherosclerotic Lesions
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Abbott Vascular
Other Study IDs: 04-800
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aproximately 1 ML blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
PROSPECT is a multi-center prospective registry of Acute Coronary Syndromes (ACS) patients with single or double vessel coronary artery disease. Approximately 700 patients with ACS will be enrolled into the study at sites in the United States and European Union.

DETAILED DESCRIPTION:
To identify in patients presenting with ACS imaging modalities and/or serologic markers of inflammation which may aid in the identification of non-flow obstructing lesions with an increased risk for future acute coronary events. This study will ascertain the prevalence and clinical significance of non-flow obstructing lesions, which subsequently result in acute coronary events - defined as vulnerable plaque. The safety of regional imaging of non-culprit lesions in ACS patients will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Acute cardiac pain, or angina equivalent, consistent with unstable angina or myocardial infarction, lasting greater than 10 minutes duration within the past 72 hours.
2. Patient must have evidence of an ACS requiring catheterization documented by the presence of any one of the following conditions:

   1. Elevated enzymes (CK-MB or troponin I or troponin T greater than upper limits of normal).
   2. ST depression of >1 mm in 2 or more contiguous leads measured at 40 ms after the J point, in the absence of left ventricular hypertrophy, bundle branch block, paced rhythms, pre-excitation or other ECG artifacts or confounding conditions.
   3. Transient ST elevation of >1 mm in 2 or more contiguous leads lasting <30 minutes (otherwise same criteria as above).
   4. ST elevation myocardial infarction with onset >24 hours previously, diagnosed with the typical triad of nitrate unresponsive chest pain lasting >30 minutes, ST elevation of >1 mm in 2 or more contiguous leads or new left bundle branch block, and rise and fall of CK-MB isoenzymes.

Key Clinical Exclusion Criteria:

1. Patient has had a documented acute ST-segment elevation myocardial infarction within the past 24 hours.
2. Known serum creatinine > 2.5 mg/dl.
3. Decompensated hypotension or heart failure requiring intubation, inotropes, intravenous diuretics or intraaortic balloon counterpulsation.
4. Patient has a known hypersensitivity, allergy or contraindication to any of the following: aspirin, heparin, clopidogrel, and ticlopidine or to contrast that cannot be adequately pre-medicated.
5. Presence of cardiac implants (i.e. implantable defibrillators); however, prior implantation of pacemaker or biventricular pacemaker is permitted.
6. Presence of cardiogenic shock.
7. Patient has a known left ventricular ejection fraction <30%.
8. Refractory ventricular arrhythmia requiring either intravenous pharmacologic treatment or defibrillator therapy (e.g. ventricular tachycardia or fibrillation).
9. Acute conduction system disease requiring temporary pacemaker insertion.
10. Patient has had a recent (within 6 months) PCI unless the patient is undergoing a staged procedure for dual vessel treatment.
11. Patient has other medical illness (i.e., cancer or congestive heart failure) or recent history of substance abuse that may cause non-compliance with the Investigational Plan, confound the data interpretation or is associated with an anticipated limited life expectancy less than one year..
12. Prior participation in this study or patient is currently enrolled in another investigational use device or drug study that has not reached its primary endpoint. If the patient is enrolled in another study that is not investigational, required visits for that trial must not interfere with the conduct of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an Acute Coronary Syndrome that require catheterization and interventional treatment of a culprit lesion(s).
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2004-10; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome variable is Non-culprit Lesion Related Major Adverse Cardiac Events; defined as the composite of cardiac death, cardiac arrest, MI, ACS, revascularization by CABG, PCI, or rehospitalization by CABG or PCI or rehospitalization for angina | Inhospital, 30 days, 180 days, 1 year and then yearly for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — Columbia University; Patrick Serruys, MD, PhD, Principal Investigator — Thoraxcenter, Erasmus University, Rotterdam, The Netherlands; Bernard de Bruyne, MD, Principal Investigator — Cardiovascular Center, OLV Hospital, Aalst, Belgium
Locations (40):
- United States (22):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Good Samaritan Hospital, San Jose, California
  - Stanford Hospital and Clinics, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - St. Vincent's Hospital and Health Care Center, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital, Kansas City, Missouri
  - Mt. Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Sisters of Charity Providence Hospitals, Columbia, South Carolina
  - St. Thomas Hospital, Nashville, Tennessee
- Belgium (2):
  - OLV-Hospital Aalst, Aalst
  - A.Z. Middleheim, Antwerp
- Skejby Sygehus, Aarhus, Denmark
- France (2):
  - CHU Jean Minjoz, Besançon
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Kerckhoff Klinik, Bad Nauheim
  - Herzzentrum Klinik für Kardiologie, Bad Oeynhausen
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
- Azienda Ospedaliera S. Orsola-Malpighi, Bologna, Italy
- Erasmus Medical Center, Rotterdam, Netherlands
- University Hospital Krakow, Krakow, Poland
- Spain (4):
  - Hospital Santa Cruz, Carnaxide
  - Hospital Clinico San Carlos, Madrid
  - University Hospital Gregorio Maranon, Madrid
  - Hospital do Meixoeiro, Vigo Pontevedra
- Sahlgrenska Sjukhuset, Gothenburg, Sweden
- University Hospital Zürich, Zurich, Switzerland
- The London Chest Hospital, London, United Kingdom

REFERENCES:
- [Result] Stone Gregg W, Lansky A.; Carlier S. et. al. A prospective, natural history study of multimodality invasive imaging to characterize vulnerable plaque: First report of the baseline findings from the PROSPECT trial. Journal of the American College of Cardiology 49(9, Suppl. B): p 19B MAR 6 2007.
- [Result] Ostuka Masato; Bruining N.; Van Pelt, N.; et.al. Three-dimensional quantification of coronary plaque burden by 64-slice computed tomography: A PROS-PECT-MSCT substudy. Journal of the American College of Cardiology 49(9, Suppl. A): p 114A MAR 6 2007
- [Result] Tanaka K; Carlier SG; Mintz GS; et.al. High risk fibroatheroma lesions are remote from the minimal lumen area site: A virtual histology IVUS analysis from the PROSPECT study AMERICAN JOURNAL OF CARDIOLOGY, 2006, V 98, N8A, P 94M-94M.
- [Derived] Gu SZ, Ahmed ME, Huang Y, Hakim D, Maynard C, Cefalo NV, Coskun AU, Costopoulos C, Maehara A, Stone GW, Stone PH, Bennett MR. Comprehensive biomechanical and anatomical atherosclerotic plaque metrics predict major adverse cardiovascular events: A new tool for clinical decision making. Atherosclerosis. 2024 Mar;390:117449. doi: 10.1016/j.atherosclerosis.2024.117449. Epub 2024 Jan 11. PMID 38262275
- [Derived] Seike F, Mintz GS, Matsumura M, Ali ZA, Liu M, Jeremias A, Ben-Yehuda O, De Bruyne B, Serruys PW, Yasuda K, Stone GW, Maehara A. Impact of Intravascular Ultrasound-Derived Lesion-Specific Virtual Fractional Flow Reserve Predicts 3-Year Outcomes of Untreated Nonculprit Lesions: The PROSPECT Study. Circ Cardiovasc Interv. 2022 Nov;15(11):851-860. doi: 10.1161/CIRCINTERVENTIONS.121.011198. Epub 2022 Nov 15. PMID 36378741
- [Derived] Farhan S, Redfors B, Maehara A, McAndrew T, Ben-Yehuda O, De Bruyne B, Mehran R, Vogel B, Giustino G, Serruys PW, Mintz GS, Stone GW. Relationship between insulin resistance, coronary plaque, and clinical outcomes in patients with acute coronary syndromes: an analysis from the PROSPECT study. Cardiovasc Diabetol. 2021 Jan 7;20(1):10. doi: 10.1186/s12933-020-01207-0. PMID 33413366
- [Derived] Farhan S, Redfors B, Maehara A, McAndrew T, Ben-Yehuda O, De Bruyne B, Mehran R, Giustino G, Kirtane AJ, Serruys PW, Mintz GS, Stone GW. Impact of Pre-Diabetes on Coronary Plaque Composition and Clinical Outcome in Patients With Acute Coronary Syndromes: An Analysis From the PROSPECT Study. JACC Cardiovasc Imaging. 2019 Apr;12(4):733-741. doi: 10.1016/j.jcmg.2017.06.023. Epub 2017 Oct 18. PMID 29055637
- [Derived] Zheng B, Mintz GS, McPherson JA, De Bruyne B, Farhat NZ, Marso SP, Serruys PW, Stone GW, Maehara A. Predictors of Plaque Rupture Within Nonculprit Fibroatheromas in Patients With Acute Coronary Syndromes: The PROSPECT Study. JACC Cardiovasc Imaging. 2015 Oct;8(10):1180-1187. doi: 10.1016/j.jcmg.2015.06.014. PMID 26481843
- [Derived] Goto K, Mintz GS, Litherland C, Lansky AJ, Weisz G, McPherson JA, De Bruyne B, Serruys PW, Stone GW, Maehara A. Lumen Measurements From Quantitative Coronary Angiography and IVUS: A PROSPECT Substudy. JACC Cardiovasc Imaging. 2016 Aug;9(8):1011-3. doi: 10.1016/j.jcmg.2015.07.006. Epub 2015 Sep 9. No abstract available. PMID 26363838
- [Derived] Xie Y, Mintz GS, Yang J, Doi H, Iniguez A, Dangas GD, Serruys PW, McPherson JA, Wennerblom B, Xu K, Weisz G, Stone GW, Maehara A. Clinical outcome of nonculprit plaque ruptures in patients with acute coronary syndrome in the PROSPECT study. JACC Cardiovasc Imaging. 2014 Apr;7(4):397-405. doi: 10.1016/j.jcmg.2013.10.010. Epub 2014 Mar 13. PMID 24631511
- [Derived] Inaba S, Mintz GS, Farhat NZ, Fajadet J, Dudek D, Marzocchi A, Templin B, Weisz G, Xu K, de Bruyne B, Serruys PW, Stone GW, Maehara A. Impact of positive and negative lesion site remodeling on clinical outcomes: insights from PROSPECT. JACC Cardiovasc Imaging. 2014 Jan;7(1):70-8. doi: 10.1016/j.jcmg.2013.10.007. PMID 24433710
- [Derived] Dohi T, Mintz GS, McPherson JA, de Bruyne B, Farhat NZ, Lansky AJ, Mehran R, Weisz G, Xu K, Stone GW, Maehara A. Non-fibroatheroma lesion phenotype and long-term clinical outcomes: a substudy analysis from the PROSPECT study. JACC Cardiovasc Imaging. 2013 Aug;6(8):908-16. doi: 10.1016/j.jcmg.2013.04.008. Epub 2013 Jul 10. PMID 23850249
- [Derived] Golinvaux N, Maehara A, Mintz GS, Lansky AJ, McPherson J, Farhat N, Marso S, de Bruyne B, Serruys PW, Templin B, Cheong WF, Aaskar R, Fahy M, Mehran R, Leon M, Stone GW. An intravascular ultrasound appraisal of atherosclerotic plaque distribution in diseased coronary arteries. Am Heart J. 2012 Apr;163(4):624-31. doi: 10.1016/j.ahj.2011.07.031. PMID 22520529
- [Derived] Sanidas EA, Mintz GS, Maehara A, Cristea E, Wennerblom B, Iniguez A, Fajadet J, Fahy M, Dressler O, Weisz G, Templin B, Zhang Z, Lansky AJ, de Bruyne B, Serruys P, Stone GW. Adverse cardiovascular events arising from atherosclerotic lesions with and without angiographic disease progression. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S95-S105. doi: 10.1016/j.jcmg.2011.08.024. PMID 22421236
- [Derived] Brener SJ, Mintz GS, Cristea E, Weisz G, Maehara A, McPherson JA, Marso SP, Farhat N, Botker HE, Dressler O, Xu K, Templin B, Zhang Z, Lansky AJ, de Bruyne B, Serruys PW, Stone GW. Characteristics and clinical significance of angiographically mild lesions in acute coronary syndromes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S86-94. doi: 10.1016/j.jcmg.2011.12.007. PMID 22421235
- [Derived] McPherson JA, Maehara A, Weisz G, Mintz GS, Cristea E, Mehran R, Foster M, Verheye S, Rabbani L, Xu K, Fahy M, Templin B, Zhang Z, Lansky AJ, de Bruyne B, Serruys PW, Stone GW. Residual plaque burden in patients with acute coronary syndromes after successful percutaneous coronary intervention. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S76-85. doi: 10.1016/j.jcmg.2012.01.005. PMID 22421234
- [Derived] Lansky AJ, Ng VG, Maehara A, Weisz G, Lerman A, Mintz GS, De Bruyne B, Farhat N, Niess G, Jankovic I, Lazar D, Xu K, Fahy M, Serruys PW, Stone GW. Gender and the extent of coronary atherosclerosis, plaque composition, and clinical outcomes in acute coronary syndromes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S62-72. doi: 10.1016/j.jcmg.2012.02.003. PMID 22421232
- [Derived] Baber U, Stone GW, Weisz G, Moreno P, Dangas G, Maehara A, Mintz GS, Cristea E, Fahy M, Xu K, Lansky AJ, Wennerblom B, Mathey DG, Templin B, Zhang Z, Serruys PW, Mehran R. Coronary plaque composition, morphology, and outcomes in patients with and without chronic kidney disease presenting with acute coronary syndromes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S53-61. doi: 10.1016/j.jcmg.2011.12.008. PMID 22421231
- [Derived] Marso SP, Mercado N, Maehara A, Weisz G, Mintz GS, McPherson J, Schiele F, Dudek D, Fahy M, Xu K, Lansky A, Templin B, Zhang Z, de Bruyne B, Serruys PW, Stone GW. Plaque composition and clinical outcomes in acute coronary syndrome patients with metabolic syndrome or diabetes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S42-52. doi: 10.1016/j.jcmg.2012.01.008. PMID 22421230
- [Derived] Papadopoulou SL, Neefjes LA, Garcia-Garcia HM, Flu WJ, Rossi A, Dharampal AS, Kitslaar PH, Mollet NR, Veldhof S, Nieman K, Stone GW, Serruys PW, Krestin GP, de Feyter PJ. Natural history of coronary atherosclerosis by multislice computed tomography. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S28-37. doi: 10.1016/j.jcmg.2012.01.009. PMID 22421228
- [Derived] Brugaletta S, Garcia-Garcia HM, Serruys PW, Maehara A, Farooq V, Mintz GS, de Bruyne B, Marso SP, Verheye S, Dudek D, Hamm CW, Farhat N, Schiele F, McPherson J, Lerman A, Moreno PR, Wennerblom B, Fahy M, Templin B, Morel MA, van Es GA, Stone GW. Relationship between palpography and virtual histology in patients with acute coronary syndromes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S19-27. doi: 10.1016/j.jcmg.2011.02.026. PMID 22421227
- [Derived] Wykrzykowska JJ, Mintz GS, Garcia-Garcia HM, Maehara A, Fahy M, Xu K, Inguez A, Fajadet J, Lansky A, Templin B, Zhang Z, de Bruyne B, Weisz G, Serruys PW, Stone GW. Longitudinal distribution of plaque burden and necrotic core-rich plaques in nonculprit lesions of patients presenting with acute coronary syndromes. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S10-8. doi: 10.1016/j.jcmg.2012.01.006. PMID 22421223
- [Derived] Maehara A, Cristea E, Mintz GS, Lansky AJ, Dressler O, Biro S, Templin B, Virmani R, de Bruyne B, Serruys PW, Stone GW. Definitions and methodology for the grayscale and radiofrequency intravascular ultrasound and coronary angiographic analyses. JACC Cardiovasc Imaging. 2012 Mar;5(3 Suppl):S1-9. doi: 10.1016/j.jcmg.2011.11.019. PMID 22421222
- [Derived] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Derived] Oviedo C, Maehara A, Mintz GS, Araki H, Choi SY, Tsujita K, Kubo T, Doi H, Templin B, Lansky AJ, Dangas G, Leon MB, Mehran R, Tahk SJ, Stone GW, Ochiai M, Moses JW. Intravascular ultrasound classification of plaque distribution in left main coronary artery bifurcations: where is the plaque really located? Circ Cardiovasc Interv. 2010 Apr;3(2):105-12. doi: 10.1161/CIRCINTERVENTIONS.109.906016. Epub 2010 Mar 2. PMID 20197513